CLINICAL TRIAL: NCT07100756
Title: Effectiveness of Implementation of Opportunistic AI-screening for Vertebral Fractures in Clinical Practice - the vertAIdo Project (Vertebral Fracture AI Detection for Better Osteoporosis Care)
Brief Title: Effectiveness of Implementation of Opportunistic AI-screening for Vertebral Fractures in Clinical Practice
Acronym: vertAIdo
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anna Spangeus, Assoc Prof MD, University Hospital, Linkoeping
Other Study IDs: vertAIdo
Record Dates: First submitted 2025-07-14; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Vertebral Fracture; Osteoporosis
Keywords: vertebral fracture; osteoporosis; computed tomography; AI
MeSH Terms: conditions — Spinal Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual care: The control cohort (usual care), representing routine care, consists of historical data from the corresponding period one year prior to the implementation of AI-based screening. In standard clinical practice, radiologists are expected to report incidental findings, including vertebral fractures. It is then the responsibility of the referring physician to act upon such findings and ensure appropriate follow-up. This includes initiating further investigation and treatment for osteoporosis in accordance with established clinical guidelines.
- AI screening aligned with FLS: In the AI cohort, an algorithm was integrated into the clinical workflow to automatically analyze CT scans of the thoracic and lumbar spine for vertebral fractures as part of opportunistic screening. Positive findings were automatically listed in the radiology PACS and subsequently reviewed and confirmed by dedicated radiologists. Confirmed fractures were referred to the Fracture Liaison Service (FLS), where a coordinator and osteoporosis specialist managed further care. Based on clinical assessment, a referral was issued to primary care, which remained responsible for continued investigation and treatment according to standard regional practice.
  Interventions: Device: AI vertebral fracture diagnostics (Flamingo)

INTERVENTIONS:
Device: AI vertebral fracture diagnostics (Flamingo) — The AI (name: Flamingo from Image Biopsy Lab, IBL, Vienna, Austria) screens thoracic and abdominal CT scans for vertebral fractures.
  Groups: AI screening aligned with FLS

SUMMARY:
The aim of this study is to evaluate clinical effectiveness and cost-effectiveness after implementing a medically approved and commercially available AI support system for opportunistic vertebral fracture screening in CT examinations within an adapted fracture care pathway (integrated care process) in clinical routine. Data will be compared to historical data (same period the previous year).

The main question it aims to answer is: Does opportunistic AI-supported vertebral fracture screening in CT examinations integrated to a fracture care pathway increase the numbers of diagnosed vertebral fractures compared to usual care?

CT scans in the clinical routine care will be opportunistically screened for vertebral fractures by the AI for 4 months. All positive findings will be confirmed by a radiologist and triaged by the FLS (Fracture Liaison Service).

DETAILED DESCRIPTION:
Objective: This study aims to compare a 4-month period during which AI support was integrated into the clinical fracture pathway (AI-cohort) with a historical cohort from the same period one year earlier (control-cohort). The prevalence of vertebral fractures on CT scans is expected to remain constant during this period.

The two cohorts include:

1. The AI-cohort where an AI algorithm was installed and integrated into the clinical workflow to automatically analyze CT images of the thoracic or lumbar spine for vertebral fractures, i.e. opportunistic screening. The AI algorithm operates on local regional servers, ensuring that no images are sent externally. A worklist of positive findings, indicating the presence of vertebral fractures, is automatically generated in the radiology PACS (Picture Archiving and Communication System). This list is reviewed and verified by dedicated radiologists to confirm the AI findings. Confirmed fractures are then linked to the fracture liaison service (FLS), where the fracture coordinator and osteoporosis specialist care for further patient management according to clinical routine, i.e. based on a medical review, writes a referral to primary care, which will be responsible for further patient investigation and treatment of osteoporosis (i.e. usual care in the region).
2. The control cohort (i.e. routine care), includes historical data from the same period the year before the AI-screening was introduced. In clinical routine, radiologists are expected to report incidental findings, such as vertebral fractures. The referring physician, who sends the referral to radiology, is then expected to act on the incidental finding of a vertebral fracture and is responsible for ensuring that the patient is managed further according to clinical routine for osteoporosis investigation and treatment.

Timeframe: Data from the AI-intervention period, spanning 4 months (20 October 2024-19 February 2025), will be analyzed. The same timeframe will be used for the historical cohort from the previous year (2023-2024).

ELIGIBILITY:
Inclusion criteria:

* abdominal or thoracic CT scans performed in clinical routine from patients living in the catchment area
* women and men
* age 50 or higher

Exclusion criteria:

-CT scans using spine-only protocol with exclusively skeletal queries

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >= 50 years, undergoing a clinical thoracic or abdominal CT-scan in at Linköping University Hospital
Sampling Method: Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Vertebral fractures (ICD coded) | Within 3 months from CT scan
  Numbers of ICD-coded vertebral fractures within 3 months from the CT scan.

SECONDARY OUTCOMES:
Reported vertebral fractures (radiology report) | Within 2 months after the CT scan
  Numbers of patients with vertebral fractures that are mentioned in the radiology report after the CT scan.
DXA screened patients | Within 12 months after the CT scan
  Numbers of patients screened with DXA (osteoporosis investigation) within 1 year after the CT scan.
Medical treatment (anti-osteoporotic) | Within 12 months after the CT scan
  Numbers of patients treated with antiosteoporotic drugs 1 year after CT scan.
Cost-effectiveness | Two time frames: Within 12 months after the CT scan and long-term using a decision-analytic model to assess outcome in 10 years
  Incremental cost per outcome compared to no AI guidance.

OTHER OUTCOMES:
Performance of AI | Baseline
  Performance (true positive, false positive, true negative and false negative) of AI detection of vertebral fractures compared to radiologist (ground truth).
  Only in the cohort "AI screening aligned with FLS"
Vertebral fractures (radiologist confirmed) | Baseline
  Numbers of vertebral fractures that are detected by AI and confirmed by radiologist in an opportunistic clinical setting. Only in the cohort "AI screening aligned with FLS".
New or worsened vertebral fractures | Baseline
  Numbers of radiologist verified vertebral fractures that were new (not previously visualised), or worsened since previous CT (minimum 3 months old). Only in the cohort "AI screening aligned with FLS"
Undiagnosed vertebral fracture | Baseline
  Numbers of old previously visualized vertebral fractures that were previously undiagnosed (ICD-code). Only in the cohort "AI screening aligned with FLS"
Untreated patients with vertebral fracture | Baseline
  Numbers of patients with vertebral fracture that were untreated at the time of the CT scan. Only in the cohort "AI screening aligned with FLS".
Patients requiring further action according to clinical triage (FLS) | 1 month
  Numbers of patients with vertebral fracture that needs further action according to the FLS. Only in the cohort "AI screening aligned with FLS".

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spångeus, Ass Prof MD, Principal Investigator — Linköpings University Hospital
Locations (1):
- Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No